CLINICAL TRIAL: NCT04329819
Title: Evaluation of the Satisfaction and the Quality of Life of Patients After Breast Reconstruction as Part of Breast Cancer. Comparison of Several Technics.
Brief Title: Satisfaction and QUality of Life After Breast REconstruction
Acronym: SQUARE
Status: Completed | Type: Observational
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Other Study IDs: ICO-2019-16
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Mammaplasty; Breast Neoplasm Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast cancer is the most common cancer in women in France in term of repercussion, 58 698 people has been diagnosed in 2017. Breast cancer is often with good prognosis. The 5 years disease-free survival rate is 87%. Surgery has a major place in breast cancer treatment. Although the conservative surgery is preferred, it stays the indication of mastectomy for nearly 30% of cases. This radical surgery is often experienced by the patient as a mutilation with the impact that this entails from a psychological point of view but also on the quality of life. Breast reconstruction allows an improvement of quality of life with a better acceptance of the body scheme and the benefits in the psychological and sexual domains. The reconstruction is an integral part of the therapeutic care; however, it is not done systematically. Indeed, in France nearly 35% of patients benefit of breast reconstruction 5 years after the mastectomy.

Nowadays, several surgical technics are available to do the reconstruction: autologous technics and the reconstruction with implants. It can be differed or immediate. The strategy of reconstruction is established in accordance with many parameters: the morphology of the breast and of the patient, the state of the thoracic wall and history of radiotherapy, comorbidities, contraindication and of course the wish of the patient. According to the used technics, the reconstruction can sometimes extend to several months, especially for the exclusive fat reshaping which needs a lot of surgery. The autologous technics seems to give a better satisfaction to the patients in an esthetical point of view but we do not have many data including the fat reshaping.

Among the tests allowing the evaluation of quality of life of patients, the Breast-Q© is a self-questionnaire validated that is specific to the breast surgery and includes a module concerning the breast reconstruction. It allows evaluating the quality of life (physical, psychosocial and sexual well-being) and the satisfaction of patients (based on cosmetic results and the care). The reconstruction module includes 116 items in its post-surgery version and is adapted to different types of reconstruction.

The objective of our project is to evaluate the quality of life and the satisfaction of patients having an immediate or differed breast reconstruction according to the technics used, with the help of the validated questionnaire Breast-Q© and the additional questionnaires.

DETAILED DESCRIPTION:
This study is retrospective and compared including exhaustively all the patients answering all inclusion criteria. The list of patients answering to all inclusion criteria will be collected with the help of the medical information department. Based on a screening on the aggregated data of the centre, the size of the sample is around 300 patients.

The medics will inform the eligible patients of the study with the help of the information note by letter. The patient will be informed of the objective if the study, the treatment of the informatics data collected during this study and the access right, the rectification, the effacement, the limit of the data treatment, the portability and opposition. This right can be done whenever to the delegate of the Data Protection.

The information letter with questionnaires will be send by post to the selected patient house. The patient responding to the questionnaires will be included in the study. In this way a part of the data will be collected directly from the answer communicated by the patient through the Breast-Q©.

Additional data will be collected in an indirect way from elements available from the informatics clinic medical file. The clinicians of the centre could be ask to complete the information.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or more
* History of mastectomy for breast cancer all types and TNM status
* Patients who beneficiated a breast reconstruction immediate or secondary finished between 01/01/2015 and 31/12/16 (not included nipples)
* Accept to answer to the questionnaire

Exclusion Criteria:

* Deceased patient
* Opposition of the patient to the data collection
* History of preventive mastectomy
* Patient who has local recurrence or metastatic cancer
* Patient under guardianship or protection of vulnerable adults

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had finished the breast reconstruction immediate or differed between 01/01/2015 and 31/12/16 whatever the technic used, following the mastectomy for breast cancer at the Institut de Cancerologie de l'Ouest, site Saint-Herblain
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Evaluate the quality of life and the satisfaction of patients who had a breast reconstruction immediate or differed according to the technics used | 2 months
  The evaluation will be done through the BREAST-Q© questionnaire (module of reconstruction and post-surgery version) The quality of life is evaluated through 6 scales (psychological and sexual well-being and also physical well-being: breast, abdomen/trunk, shoulder/back). The satisfaction is evaluated with 9 scales (satisfaction of breast, nipples, abdomen, back and treatment: information received, surgeon, medical team and administrative staff).
  There is no global score for BREAST- Q©. Each scale is independent and converted from 0 to 100. A high score means a better satisfaction of quality of life.

SECONDARY OUTCOMES:
Describe the practices in term of breast reconstruction in the Institut de Cancerologie de l'Ouest-site Saint-Herblain. | 2 months
  The frequency of different technics used in the ICO site Saint-Herblain will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Victoire BRILLAUD-MEFLAH, Principal Investigator — Institut de Cancerologie de l'Ouest
Locations (1):
- Institut de Cancerologie de l'Ouest, Saint-Herblain, France